CLINICAL TRIAL: NCT01484457
Title: Controlled Insulin Delivery: Combining Technology With Treatment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Schneider Children's Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JDRF 22-2009-796
Record Dates: First submitted 2011-11-15; First posted 2011-12-02 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus; Closed Loop; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Closed-loop control system (Experimental): The objective of this study is to automate glucose control in subjects with type 1 diabetes using a computer control algorithm in a controlled in-clinic research setting.
  The controller will be evaluated under two conditions:
  1. restoring euglycemia (80-140 mg/dL) when the controller is initiated during a period when the subject's glucose is above the euglycemic range;
  2. restoring euglycemia (80-140 mg/dL) when the controller is challenged with a small unannounced meal (~25 g CHO).
  Interventions: Device: Closed-loop session

INTERVENTIONS:
Device: Closed-loop session — Subjects will arrive fasting at 7am unless needed for hypoglycemia (glucose < 70 mg/dL) and no extra bolus insulin after 3am. An IV catheter will be inserted for blood samples and for IV administration of glucose if necessary. Blood samples will be analyzed for glucose by YSI 2300Stat every 30 minutes.
  Breakfast consisting of 25g of CHO will be eaten at 7:30 am and the subject will bolus for this amount of CHO. The controller is switched "on" on the down slope of the meal response, and the subject is brought to a basal steady-state by the controller. Target blood glucose is 110 ± 30-mg/dL.
  After approximately 3 hours a small lunch will be eaten consisting of 25g of CHO (unannounced meal challenge). The subject will be monitored until blood glucose returns to euglycemia.
  Other Names: Closed-loop Artificial Pancreas Device

SUMMARY:
Hypothesis: Closed-loop control systems for an artificial pancreas using multi-parametric model predictive control can be developed and evaluated safely in patients with Type 1 Diabetes Mellitus (T1DM) to control blood glucose concentrations.

This study seeks to combine real-time continuous glucose sensing with automated insulin delivery in a closed-loop system that will achieve euglycemia in patients with T1DM. The end result of this line of research will be an artificial pancreas that will provide around-the-clock glucose regulation through controlled insulin delivery in response to detected patterns of change in glucose levels.

DETAILED DESCRIPTION:
The goal of the JDRF Artificial Pancreas Project is to produce an autonomous artificial pancreas that can safely and effectively regulate glycemia in people with type 1 diabetes mellitus. In our work, this fully automated closed-loop system combines a subcutaneous continuous glucose monitor (CGM) and a continuous subcutaneous insulin infusion (CSII) pump with a sophisticated control algorithm. This is a proof-of-concept study to demonstrate that the controller could bring the patient back to a relatively normal glucose concentration after an unannounced meal and from mild hyperglycemia. Once the system is initiated, all insulin delivery is calculated automatically. There was no outside intervention either by the subject or medical personnel. An artificial pancreas system that aims at replicating normal beta-cell function by using the subcutaneous-subcutaneous (sc-sc) route needs to address inherent delays in both glucose sensing and insulin delivery. Our strategic approach is that a closed-loop system should operate safely without any knowledge of meals or other disturbances. We have developed the Artificial Pancreas System (APS©) and used it to clinically evaluate a control strategy that allows efficient glycemic control without any a priori meal information. The Artificial Pancreas device uses the Artificial Pancreas System (APS©) platform with the OmniPod insulin pump, the DexCom SEVEN PLUS CGM and a multi-parametric model predictive control algorithm (mpMPC) with an insulin-on-board (IOB) safety constraint.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the consent form
2. Type 1 diabetes for at least 1 year prior to the study
3. Using continuous subcutaneous insulin infusion pump
4. Above 21 years of age
5. Willing to follow the study requirements

Exclusion Criteria:

1. Allergy to the sensor or to one of its components
2. Psychiatric disorders
3. Reported diabetic ketoacidosis within last 3 months
4. Abnormal liver function (Transaminase > 2 times the upper limit of normal)
5. Heart failure
6. Any carcinogenic disease
7. Any other chronic abnormality
8. Unwilling to perform or to follow the research protocol
9. Participation in any other study concurrent with the proposed study
10. Creatinine concentration above the upper limit of normal for age and sex
11. Active coronary artery disease
12. Active gastroparesis
13. History of uncontrolled seizures
14. Pregnancy
15. Untreated adrenal insufficiency
16. Hypokalemia
17. Uncontrolled thyroid disease.
18. Condition, which in the opinion of the investigator, would interfere with patient safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Restoration of Euglycemia | 12 hours
  The primary endpoint of this pilot study is successful restoration of euglycemia from the two perturbed conditions using closed loop control with minimal hypo- and hyperglycemia exposure. The first condition involves restoration of euglycemia when the subject is in a hyperglycemic state. The second condition involves restoration of euglycemia following consumption of a meal containing 25g CHO with no insulin bolus. The patients will be followed for the duration of the 12 hour study.

SECONDARY OUTCOMES:
Average percent-of-time-in-range (80 - 180 mg/dL) | 12 hours
  All reported blood glucose values per both CGM and YSI ware analyzed for average percent-of-time-in-range (80 - 180 mg/dL). The participants will be followed for the duration of the 12 hour study.

CONTACTS AND LOCATIONS:
Overall Officials: Lois Jovanovic, M.D., Principal Investigator — Sansum Diabetes Research Institute
Locations (2):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

REFERENCES:
- [Background] Basu R, Di Camillo B, Toffolo G, Basu A, Shah P, Vella A, Rizza R, Cobelli C. Use of a novel triple-tracer approach to assess postprandial glucose metabolism. Am J Physiol Endocrinol Metab. 2003 Jan;284(1):E55-69. doi: 10.1152/ajpendo.00190.2001. PMID 12485809
- [Background] Bellazzi R, Arcelloni M, Bensa G, Blankenfeld H, Brugues E, Carson E, Cobelli C, Cramp D, D'Annunzio G, De Cata P, De Leiva A, Deutsch T, Fratino P, Gazzaruso C, Garcia A, Gergely T, Gomez E, Harvey F, Ferrari P, Hernando E, Boulos MK, Larizza C, Ludekke H, Maran A, Nucci G, Pennati C, Ramat S, Roudsari A, Rigla M, Stefanelli M. Design, methods, and evaluation directions of a multi-access service for the management of diabetes mellitus patients. Diabetes Technol Ther. 2003;5(4):621-9. doi: 10.1089/152091503322250640. PMID 14511417
- [Background] Bellazzi R, Nucci G, Cobelli C. The subcutaneous route to insulin-dependent diabetes therapy. IEEE Eng Med Biol Mag. 2001 Jan-Feb;20(1):54-64. doi: 10.1109/51.897828. No abstract available. PMID 11211661
- [Background] Bequette BW. A critical assessment of algorithms and challenges in the development of a closed-loop artificial pancreas. Diabetes Technol Ther. 2005 Feb;7(1):28-47. doi: 10.1089/dia.2005.7.28. PMID 15738702
- [Background] Bevier WC, Zisser H, Palerm CC, Finan DA, Seborg DE, Doyle FJ, Wollitzer AO, Jovanovic L. Calculating the insulin to carbohydrate ratio using the hyperinsulinaemic-euglycaemic clamp-a novel use for a proven technique. Diabetes Metab Res Rev. 2007 Sep;23(6):472-8. doi: 10.1002/dmrr.727. PMID 17315240
- [Background] Bode BW. Clinical utility of the continuous glucose monitoring system. Diabetes Technol Ther. 2000;2 Suppl 1:S35-41. doi: 10.1089/15209150050214104. No abstract available. PMID 11469630
- [Background] Bode BW, Gross TM, Thornton KR, Mastrototaro JJ. Continuous glucose monitoring used to adjust diabetes therapy improves glycosylated hemoglobin: a pilot study. Diabetes Res Clin Pract. 1999 Dec;46(3):183-90. doi: 10.1016/s0168-8227(99)00113-8. PMID 10624783
- [Background] Bode BW, Hirsch IB. Using the continuous glucose monitoring system to improve the management of type 1 diabetes. Diabetes Technol Ther. 2000;2 Suppl 1:S43-8. doi: 10.1089/15209150050214113. No abstract available. PMID 11469631
- [Background] Broekhuyse HM, Nelson JD, Zinman B, Albisser AM. Comparison of algorithms for the closed-loop control of blood glucose using the artificial beta cell. IEEE Trans Biomed Eng. 1981 Oct;28(10):678-87. doi: 10.1109/tbme.1981.324661. No abstract available. PMID 7033107
- [Background] Chanoch LH, Jovanovic L, Peterson CM. The evaluation of a pocket computer as an aid to insulin dose determination by patients. Diabetes Care. 1985 Mar-Apr;8(2):172-6. doi: 10.2337/diacare.8.2.172. PMID 3838930
- [Background] Dalla Man C, Caumo A, Basu R, Rizza R, Toffolo G, Cobelli C. Measurement of selective effect of insulin on glucose disposal from labeled glucose oral test minimal model. Am J Physiol Endocrinol Metab. 2005 Nov;289(5):E909-14. doi: 10.1152/ajpendo.00299.2004. Epub 2005 Jun 21. PMID 15972269
- [Background] Dassau E, Palerm CC, Zisser H, Buckingham BA, Jovanovic L, Doyle FJ. In silico evaluation platform for artificial pancreatic beta-cell development--a dynamic simulator for closed-loop control with hardware-in-the-loop. Diabetes Technol Ther. 2009 Mar;11(3):187-94. doi: 10.1089/dia.2008.0055. PMID 19191486
- [Background] Dassau E, Zisser H, C Palerm C, A Buckingham B, Jovanovic L, J Doyle F 3rd. Modular artificial beta-cell system: a prototype for clinical research. J Diabetes Sci Technol. 2008 Sep;2(5):863-72. doi: 10.1177/193229680800200518. PMID 19885271
- [Background] Diabetes Research in Children Network (DirecNet) Study Group; Buckingham B, Beck RW, Tamborlane WV, Xing D, Kollman C, Fiallo-Scharer R, Mauras N, Ruedy KJ, Tansey M, Weinzimer SA, Wysocki T. Continuous glucose monitoring in children with type 1 diabetes. J Pediatr. 2007 Oct;151(4):388-93, 393.e1-2. doi: 10.1016/j.jpeds.2007.03.047. Epub 2007 Aug 24. PMID 17889075
- [Background] Dua P, Doyle FJ 3rd, Pistikopoulos EN. Model-based blood glucose control for Type 1 diabetes via parametric programming. IEEE Trans Biomed Eng. 2006 Aug;53(8):1478-91. doi: 10.1109/TBME.2006.878075. PMID 16916082
- [Background] Garg S, Zisser H, Schwartz S, Bailey T, Kaplan R, Ellis S, Jovanovic L. Improvement in glycemic excursions with a transcutaneous, real-time continuous glucose sensor: a randomized controlled trial. Diabetes Care. 2006 Jan;29(1):44-50. doi: 10.2337/diacare.29.01.06.dc05-1686. PMID 16373894
- [Background] Hovorka R, Chassin LJ, Wilinska ME, Canonico V, Akwi JA, Federici MO, Massi-Benedetti M, Hutzli I, Zaugg C, Kaufmann H, Both M, Vering T, Schaller HC, Schaupp L, Bodenlenz M, Pieber TR. Closing the loop: the adicol experience. Diabetes Technol Ther. 2004 Jun;6(3):307-18. doi: 10.1089/152091504774197990. PMID 15198833
- [Background] Hovorka R, Shojaee-Moradie F, Carroll PV, Chassin LJ, Gowrie IJ, Jackson NC, Tudor RS, Umpleby AM, Jones RH. Partitioning glucose distribution/transport, disposal, and endogenous production during IVGTT. Am J Physiol Endocrinol Metab. 2002 May;282(5):E992-1007. doi: 10.1152/ajpendo.00304.2001. PMID 11934663
- [Background] Jeha GS, Karaviti LP, Anderson B, Smith EO, Donaldson S, McGirk TS, Haymond MW. Insulin pump therapy in preschool children with type 1 diabetes mellitus improves glycemic control and decreases glucose excursions and the risk of hypoglycemia. Diabetes Technol Ther. 2005 Dec;7(6):876-84. doi: 10.1089/dia.2005.7.876. PMID 16386093
- [Background] Jones SM, Quarry JL, Caldwell-McMillan M, Mauger DT, Gabbay RA. Optimal insulin pump dosing and postprandial glycemia following a pizza meal using the continuous glucose monitoring system. Diabetes Technol Ther. 2005 Apr;7(2):233-40. doi: 10.1089/dia.2005.7.233. PMID 15857224
- [Background] Jovanovic L. Role of diet and insulin treatment of diabetes in pregnancy. Clin Obstet Gynecol. 2000 Mar;43(1):46-55. doi: 10.1097/00003081-200003000-00005. No abstract available. PMID 10694987
- [Background] Kan S, Onodera H, Furutani E, Aung T, Araki M, Nishimura H, Maetani S, Imamura M. Novel control system for blood glucose using a model predictive method. ASAIO J. 2000 Nov-Dec;46(6):657-62. doi: 10.1097/00002480-200011000-00004. PMID 11110261
- [Background] Kaufman FR. Searching for glycemic control in pediatric type 1 diabetes: A long way to go. J Pediatr. 2001 Aug;139(2):174-6. doi: 10.1067/mpd.2001.117573. No abstract available. PMID 11487739
- [Background] Klonoff DC. Continuous glucose monitoring: roadmap for 21st century diabetes therapy. Diabetes Care. 2005 May;28(5):1231-9. doi: 10.2337/diacare.28.5.1231. No abstract available. PMID 15855600
- [Background] Klonoff DC. A review of continuous glucose monitoring technology. Diabetes Technol Ther. 2005 Oct;7(5):770-5. doi: 10.1089/dia.2005.7.770. No abstract available. PMID 16241880
- [Background] Kovatchev BP, Cox DJ, Gonder-Frederick LA, Young-Hyman D, Schlundt D, Clarke W. Assessment of risk for severe hypoglycemia among adults with IDDM: validation of the low blood glucose index. Diabetes Care. 1998 Nov;21(11):1870-5. doi: 10.2337/diacare.21.11.1870. PMID 9802735
- [Background] Lehmann ED, Deutsch T. A physiological model of glucose-insulin interaction in type 1 diabetes mellitus. J Biomed Eng. 1992 May;14(3):235-42. doi: 10.1016/0141-5425(92)90058-s. PMID 1588781
- [Background] Lehmann ED, Deutsch T. Compartmental models for glycaemic prediction and decision-support in clinical diabetes care: promise and reality. Comput Methods Programs Biomed. 1998 May;56(2):193-204. doi: 10.1016/s0169-2607(98)00025-x. PMID 9700433
- [Background] Livesey G, Wilson PD, Dainty JR, Brown JC, Faulks RM, Roe MA, Newman TA, Eagles J, Mellon FA, Greenwood RH. Simultaneous time-varying systemic appearance of oral and hepatic glucose in adults monitored with stable isotopes. Am J Physiol. 1998 Oct;275(4):E717-28. doi: 10.1152/ajpendo.1998.275.4.E717. PMID 9755093
- [Background] Ludvigsson J, Hanas R. Continuous subcutaneous glucose monitoring improved metabolic control in pediatric patients with type 1 diabetes: a controlled crossover study. Pediatrics. 2003 May;111(5 Pt 1):933-8. doi: 10.1542/peds.111.5.933. PMID 12728068
- [Background] Magni L, Raimondo DM, Man CD, Breton M, Patek S, Nicolao GD, Cobelli C, Kovatchev BP. Evaluating the efficacy of closed-loop glucose regulation via control-variability grid analysis. J Diabetes Sci Technol. 2008 Jul;2(4):630-5. doi: 10.1177/193229680800200414. PMID 19885239
- [Background] Matsuo Y, Shimoda S, Sakakida M, Nishida K, Sekigami T, Ichimori S, Ichinose K, Shichiri M, Araki E. Strict glycemic control in diabetic dogs with closed-loop intraperitoneal insulin infusion algorithm designed for an artificial endocrine pancreas. J Artif Organs. 2003;6(1):55-63. doi: 10.1007/s100470300009. PMID 14598126
- [Background] Mauras N, Beck RW, Ruedy KJ, Kollman C, Tamborlane WV, Chase HP, Buckingham BA, Tsalikian E, Weinzimer S, Booth AD, Xing D; Diabetes Research in Children Network (DirecNet) Accuracy Study. Lack of accuracy of continuous glucose sensors in healthy, nondiabetic children: results of the Diabetes Research in Children Network (DirecNet) accuracy study. J Pediatr. 2004 Jun;144(6):770-5. doi: 10.1016/j.jpeds.2004.03.042. PMID 15192625
- [Background] Owens C, Zisser H, Jovanovic L, Srinivasan B, Bonvin D, Doyle FJ 3rd. Run-to-run control of blood glucose concentrations for people with Type 1 diabetes mellitus. IEEE Trans Biomed Eng. 2006 Jun;53(6):996-1005. doi: 10.1109/TBME.2006.872818. PMID 16761826
- [Background] Palerm CC, Zisser H, Bevier WC, Jovanovic L, Doyle FJ 3rd. Prandial insulin dosing using run-to-run control: application of clinical data and medical expertise to define a suitable performance metric. Diabetes Care. 2007 May;30(5):1131-6. doi: 10.2337/dc06-2115. Epub 2007 Feb 15. PMID 17303792
- [Background] Palerm CC, Zisser H, Jovanovic L, Doyle FJ 3rd. A Run-to-Run Control Strategy to Adjust Basal Insulin Infusion Rates in Type 1 Diabetes. J Process Control. 2008;18(3-4):258-265. doi: 10.1016/j.jprocont.2007.07.010. PMID 18709180
- [Background] Parker RS, Doyle FJ 3rd, Peppas NA. A model-based algorithm for blood glucose control in type I diabetic patients. IEEE Trans Biomed Eng. 1999 Feb;46(2):148-57. doi: 10.1109/10.740877. PMID 9932336
- [Background] Parker RS, Doyle FJ 3rd, Peppas NA. The intravenous route to blood glucose control. IEEE Eng Med Biol Mag. 2001 Jan-Feb;20(1):65-73. doi: 10.1109/51.897829. No abstract available. PMID 11211662
- [Background] Peterson CM, Jones RL, Drexler AJ, Jovanovic LB. A randomized comparative crossover evaluation of glucose monitoring technologies. Diabetes Res. 1984 Nov;1(4):195-9. PMID 6529891
- [Background] Peterson CM, Jovanovic L, Chanoch LH. Randomized trial of computer-assisted insulin delivery in patients with type I diabetes beginning pump therapy. Am J Med. 1986 Jul;81(1):69-72. doi: 10.1016/0002-9343(86)90184-1. PMID 3524226
- [Background] Palerm CC, Rodriguez-Fernandez M, Bevier WC, Zisser H, Banga JR, Jovanovic L, Doyle FJ 3rd. Robust parameter estimation in a model for glucose kinetics in type 1 diabetes subjects. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:319-22. doi: 10.1109/IEMBS.2006.260045. PMID 17946395
- [Background] Shimoda S, Nishida K, Sakakida M, Konno Y, Ichinose K, Uehara M, Nowak T, Shichiri M. Closed-loop subcutaneous insulin infusion algorithm with a short-acting insulin analog for long-term clinical application of a wearable artificial endocrine pancreas. Front Med Biol Eng. 1997;8(3):197-211. PMID 9444512
- [Background] Steil GM, Clark B, Kanderian S, Rebrin K. Modeling insulin action for development of a closed-loop artificial pancreas. Diabetes Technol Ther. 2005 Feb;7(1):94-108. doi: 10.1089/dia.2005.7.94. PMID 15738707
- [Background] Steil GM, Panteleon AE, Rebrin K. Closed-loop insulin delivery-the path to physiological glucose control. Adv Drug Deliv Rev. 2004 Feb 10;56(2):125-44. doi: 10.1016/j.addr.2003.08.011. PMID 14741112
- [Background] Tanenberg R, Bode B, Lane W, Levetan C, Mestman J, Harmel AP, Tobian J, Gross T, Mastrototaro J. Use of the Continuous Glucose Monitoring System to guide therapy in patients with insulin-treated diabetes: a randomized controlled trial. Mayo Clin Proc. 2004 Dec;79(12):1521-6. doi: 10.4065/79.12.1521. PMID 15595336
- [Background] Trajanoski Z, Wach P. Neural predictive controller for insulin delivery using the subcutaneous route. IEEE Trans Biomed Eng. 1998 Sep;45(9):1122-34. doi: 10.1109/10.709556. PMID 9735562
- [Background] Wilinska ME, Chassin LJ, Schaller HC, Schaupp L, Pieber TR, Hovorka R. Insulin kinetics in type-I diabetes: continuous and bolus delivery of rapid acting insulin. IEEE Trans Biomed Eng. 2005 Jan;52(1):3-12. doi: 10.1109/TBME.2004.839639. PMID 15651559
- [Background] Zisser H, Jovanovic L, Doyle F 3rd, Ospina P, Owens C. Run-to-run control of meal-related insulin dosing. Diabetes Technol Ther. 2005 Feb;7(1):48-57. doi: 10.1089/dia.2005.7.48. PMID 15738703
- [Background] Zisser H, Robinson L, Bevier W, Dassau E, Ellingsen C, Doyle FJ, Jovanovic L. Bolus calculator: a review of four "smart" insulin pumps. Diabetes Technol Ther. 2008 Dec;10(6):441-4. doi: 10.1089/dia.2007.0284. PMID 19049372
- [Background] Zisser HC, Bevier WC, Jovanovic L. Restoring euglycemia in the basal state using continuous glucose monitoring in subjects with type 1 diabetes mellitus. Diabetes Technol Ther. 2007 Dec;9(6):509-15. doi: 10.1089/dia.2007.0220. PMID 18034605